CLINICAL TRIAL: NCT05296486
Title: Influence of Different Tamponade Eyes on IOL-capsular Complex After Cataract Surgery Combined With Vitrectomy
Brief Title: Influence of Different Tamponade Eyes on IOL-capsular Complex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IOL with different tamponade
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Cataract; Vitreoretinal Abnormality
Keywords: Various Types of intravitreal tamponade materials
MeSH Terms: conditions — Cataract | interventions — Vitrectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- phacovitrectomy surgery with silicone oil tamponade (Experimental): patients who had phacovitrectomy surgery with silicone oil tamponade.The patients diagnosed cataract The patients' ages are over 50.
  Interventions: Procedure: phacovitrectomy surgery with silicone oil tamponade
- phacovitrectomy surgery with gas tamponade (Experimental): patients who had phacovitrectomy surgery with gas tamponade.The patients diagnosed cataract The patients' ages are over 50.
  Interventions: Procedure: phacovitrectomy surgery with gas tamponade
- phacovitrectomy surgery with balanced saline solution tamponade (Experimental): patients who had phacovitrectomy surgery with balanced saline solution tamponade.The patients diagnosed cataract The patients' ages are over 50.
  Interventions: Procedure: phacovitrectomy surgery with balanced saline solution tamponade
- phacoemulsifacation surgery without vitrectomy (Experimental): patients who had phacoemulsifacation surgery without vitrectomy.The patients diagnosed cataract The patients' ages are over 50.
  Interventions: Procedure: phacoemulsifacation surgery without vitrectomy

INTERVENTIONS:
Procedure: phacovitrectomy surgery with silicone oil tamponade — Patients in this study will receive phacovitrectomy surgery with silicone oil tamponade.
  Arms: phacovitrectomy surgery with silicone oil tamponade
Procedure: phacovitrectomy surgery with gas tamponade — Patients in this study will receive phacovitrectomy surgery with gas tamponade
  Arms: phacovitrectomy surgery with gas tamponade
Procedure: phacovitrectomy surgery with balanced saline solution tamponade — Patients in this study will receive phacovitrectomy surgery with balanced saline solution tamponade
  Arms: phacovitrectomy surgery with balanced saline solution tamponade
Procedure: phacoemulsifacation surgery without vitrectomy — Patients in this study will receive phacoemulsifacation surgery without vitrectomy.
  Arms: phacoemulsifacation surgery without vitrectomy

SUMMARY:
Cataract and vitreoretinal diseases often occur simultaneously or cataract is a predictable consequence of vitreoretinal surgery.A combined surgery called phacovitrectomy, has been proved to be comparably safe and effective compared with vitrectomy alone. For fundus surgeons, silicone oil（SO）,gas and balanced saline solution are frequently-used intravitreal tamponade mediums for retinal repair after vitrectomy. There are many factors that may affect how the lens changes position after the operation including the different intravitreal tamponade materials and different IOL types. This study was designed to evaluate the differences of IOL position and capsule bending between Silicone oil filled eyes，gas filled eyes, balanced saline solution filled eyes and normal eyes.

The IOL-capsular complex is formed after cataract surgery and intraocular lens (IOL) implantation. Early postoperative mechanical wrapping of the anterior and posterior capsules plays a significant role in preventing IOL decentration and tilt, as well as formation of the IOL-capsular complex which reduces the incidence of posterior cataract opacity.

Although up to 2-3 degree tilt and a 0.2-0.3 mm decentration are common and clinically unnoticed, larger extent of tilt and decentration has a negative impact on the optical performance. IOL decentration ≥ 0.4 mm or/and IOL tilt ≥7degree were considered clinically significant because of poor post-surgery visual quality.

Currently, there is no literature guidance to compare the results of phacovitrectomy combined various types of intravitreal tamponade materials in patients using CASIA2. The novel anterior segment optical coherence tomography (AS-OCT) device, CASIA2 can evaluate the IOL capsule bending and the lens position after cataract surgery. Also, CASIA2 can be used to documented the dynamic changes of IOL-capsular complex after surgery.

DETAILED DESCRIPTION:
Cataract and vitreoretinal diseases often occur simultaneously or cataract is a predictable consequence of vitreoretinal surgery. Although the optimal treatment for patients with both vitreoretinal and cataract disease is still a matter of debate, a combined surgery called phacovitrectomy, has been proved to be comparably safe and effective compared with vitrectomy alone. For fundus surgeons, silicone oil（SO）,gas and balanced saline solution are frequently-used intravitreal tamponade mediums for retinal repair after vitrectomy. As a biochemically inert polymer, SO is widely used in vitreoretinal surgery and was considered to be well-tolerated and not threatening to retinal physiology. The gases in therapeutic use ([SF6], [C2F6], or [C3F8]) may be mixed with air in vitrectomy or used as 100% gas in pneumatic retinopexy. There are many factors that may affect how the lens changes position after the operation including the different intravitreal tamponade materials and different IOL types. This study was designed to evaluate the differences of IOL position and capsule bending between Silicone oil filled eyes，gas filled eyes, balanced saline solution filled eyes and normal eyes.

The IOL-capsular complex is formed after cataract surgery and intraocular lens (IOL) implantation. Early postoperative mechanical wrapping of the anterior and posterior capsules plays a significant role in preventing IOL decentration and tilt, as well as formation of the IOL-capsular complex which reduces the incidence of posterior cataract opacity.

Although up to 2-3 degree tilt and a 0.2-0.3 mm decentration are common and clinically unnoticed, larger extent of tilt and decentration has a negative impact on the optical performance. IOL decentration ≥ 0.4 mm or/and IOL tilt ≥7degree were considered clinically significant because of poor post-surgery visual quality.

Currently, there is no literature guidance to compare the results of phacovitrectomy combined various types of intravitreal tamponade materials in patients using CASIA2. The novel anterior segment optical coherence tomography (AS-OCT) device, CASIA2 can evaluate the IOL capsule bending and the lens position after cataract surgery. Also, CASIA2 can be used to documented the dynamic changes of IOL-capsular complex after surgery.

ELIGIBILITY:
Inclusion Criteria:

* The patients are diagnosed age related cataract or complicated cataract with or without vitreoretinal diseases
* The patients' age over 50 years old
* The patients plan to receive cataract surgery with or without vitrectomy in Eye hospital of Wenzhou Medical University
* The dilated pupils are over 7mm
* Patients are willing and able to complete the follow-ups.

Exclusion Criteria:

* Patients with other type of cataract
* Patients have severe complications in the surgery and after surgery
* Patients have other severe diseases of eyes

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The position of IOL | The 1st day after surgery
  Evaluation of the position of IOL through tilt, decentration，rotation and the process of capsule bending using CAISA2（The novel anterior segment optical coherence tomography (AS-OCT) device）
The position of IOL | The 1st week after surgery
  Evaluation of the position of IOL through tilt, decentration，rotation and the process of capsule bending using CAISA2（The novel anterior segment optical coherence tomography (AS-OCT) device）
The position of IOL | The 1st month after surgery
  Evaluation of the position of IOL through tilt, decentration，rotation and the process of capsule bending using CAISA2（The novel anterior segment optical coherence tomography (AS-OCT) device）
The position of IOL | The 3rd month after surgery
  Evaluation of the position of IOL through tilt, decentration，rotation and the process of capsule bending using CAISA2（The novel anterior segment optical coherence tomography (AS-OCT) device）

CONTACTS AND LOCATIONS:
Overall Officials: Yune Zhao, Study Director — Ophthalmology and Optometry Hospital

IPD SHARING:
Plan to Share IPD: No